CLINICAL TRIAL: NCT02764645
Title: A Study to Collect Additional Information Related to the Performance of the CARDIOGARD Cannula
Brief Title: Performance of the CARDIOGARD Cannula
Acronym: GECG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: CardioGard Medical Ltd. (Industry)
Responsible Party: Principal Investigator, Gil Bolotin MD, Professor, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLNG100 Full Protocol
Record Dates: First submitted 2016-03-22; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Heart Valve Diseases; Coronary Artery Disease
Keywords: Cardiopulmonary Bypass
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CardioGard group (Experimental): Patients in whom the CardioGard Cannula will be used, while In these patients there would be a measurement of the gaseous emboli in two points: 1. The aortic vent.
  2. The suction cannula of the 'Cardiogard cannula'.
  Interventions: Device: CardioGard Cannula
- Control group (Active Comparator): Patients in whom a 22Fr curved Cannula will be used, while In these patients there would be a measurement of the gaseous emboli in the aortic vent alone.
  Interventions: Device: 22Fr curved Cannula

INTERVENTIONS:
Device: CardioGard Cannula — CardioGard Cannula is a specially designed arterial (aortic) cannula for use in cardiac surgery for the purpose of removal of gaseous and solid embolic material emanating during the CPB procedure.
  The CardioGard cannula is a double lumen cannula where the primary lumen provides blood from the heart-lung machine similar to ordinary cannulas and the secondary lumen performs suction of blood and embolic matter away from the aortic arch and back to the cardiopulmonary bypass machine for filtration.
  Arms: CardioGard group
Device: 22Fr curved Cannula — arterial cannula for use in cardiac surgery
  Arms: Control group

SUMMARY:
This is a single center, prospective study:

The 'CardioGard Cannula' Gaseous emboli capture results - shows an improvement from the control group.

DETAILED DESCRIPTION:
Patients referred for CPB procedure will be offered to participate in the study. Patients will be asked to sign an informed consent form (ICF), prior to performing any study related procedures.

The point of enrollment is the time at which a patient signs and dates the ICF. Following enrollment, the patient will undergo screening evaluation (including Neurological assessment) to determine eligibility. Screening failures will be identified on a screening log. Patients who are found to meet all inclusion criteria and none of the exclusion criteria will compose the evaluable cohort of the study. Screening failure subjects will not be counted as part of the target patient sample size nor will they be included in the analysis.

Patients in the randomized phase will have surgery with the CardioGard Cannula or comparator cannulae and will remain blinded to their group assignment through the 30 days follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient indicated for first-time non-emergent procedure under cardiopulmonary bypass which is expected to last up to 6 hours.
2. Patient undergoing an elective isolated coronary artery bypass surgery (CABG), or an elective isolated aortic/mitral valve replacement (AVR/MVR) or an elective combined aortic/mitral valve replacement (AVR/MVR) with coronary artery bypass surgery (CABG).
3. The patient is >50 and <85 years of age.
4. The patient's body weight is compatible with blood net flow of 4 - 5 [l/min].
5. Patient with left ventricular ejection fraction >30% as assessed by either echocardiography, angiography or by radio nuclear assessment (MUGA)
6. The patient is willing to participate as evidenced by signing the written informed consent.
7. Male or non-pregnant female patient (Note: Females of child bearing potential must have a negative pregnancy test)

Exclusion Criteria:

1. Patient with abnormal clotting mechanism: PT 60%, PTT>2 the normal.
2. Patient with an aortic trauma.
3. Patient contraindicated for open heart surgery under bypass machine.
4. Patient undergoing a re-do procedure.
5. Patient intended for an operation performed using minimally invasive surgical techniques (e.g., mini-sternotomy)
6. Patient with pathologies which affect his/her neurological condition.
7. Patient in whom emergency operation is required.
8. Patient with a known allergy to Heparin
9. Patient with major co-morbid condition(s) that could limit the patient's ability to participate in the study, or impact the scientific integrity of the study, including but not limited to:

   * previous stroke
   * critical preoperative state
   * poor ventricular function
   * severe pulmonary hypertension [19]
   * Atheroembolism
   * history of cardiac failure [20]
10. Current use of drugs that might result in high surgical risk or significant postoperative complication.
11. Psychological instability, inappropriate attitude or motivation.
12. Patients with life threatening debilitating disease other than cardiac.
13. Subjects currently enrolled in another investigational device or drug trial that has not completed the primary end point or that clinically interferes with the current study endpoints.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The 'CardioGard Cannula' Gaseous emboli capturing ability | 36 months
  The gaseous emboli capturing ability of the cardiogard cannula will be evaluated using a bubbles counter. .

SECONDARY OUTCOMES:
The amount of emboli particles which evacuated from the cardiopulmonarybypass machine by the CardioGard Cannula | 36 months
  Using the suction feature, External filters will be analyzed in order to recover particulate matter.
The Neurological effect of reducing gaseous emboli from the heart during cardiac surgery. | 36 months
  The ability of the Cardiogard cannula will be evaluated using Neurological questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Gil - Bolotin, Prof., Principal Investigator — Head of the Cardiac Surgery Department, Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Yes
The data of this research would be published as an article and will include all the relevant clinical outcomes related to the effect of gaseous emboli.